CLINICAL TRIAL: NCT01873742
Title: The STIC Online Feedback System in Psychotherapy Process-outcome Research: A Multi-site, Multi-modality, International RCT-study.
Brief Title: The STIC Norway RCT Study: Using Feedback in Psychotherapy.
Acronym: STICNorway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Principal Investigator, Terje Tilden, PhD, Terje Tilden, PhD, Modum Bad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Tilden; 2012/2/0275 (Other: Rådet for psykisk helse, Norway)
Record Dates: First submitted 2013-02-21; First posted 2013-06-10 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Psychological Feedback
Keywords: Psychotherapy feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The use of STIC feedback system (Experimental): This will constitute the experimental condition, using of STIC feedback system.
  Interventions: Other: STIC feedback system
- Treatment as usual (Experimental): This condition will not include the use of the STIC feedback system.
  Interventions: Other: STIC feedback system

INTERVENTIONS:
Other: STIC feedback system — This condition includes the use of the STIC feedback system.

SUMMARY:
Feedback in psychotherapy involves clients monitoring therapy process and progress, and on a frequent basis clients register these data into online questionnaires. These data are then fed back to the therapist, hence informing about the process and progress in therapy. This information can be shared with the client, something that may enhance the client involvement in evaluating and planning of the therapy. The same data can be used for research purpose. This randomized controlled multicenter study within Norwegian couple and family contexts will explore the effects of feedback in natural settings, and it collaborates closely with a similar American study in Chicago/Evanston, Ill.

DETAILED DESCRIPTION:
The improvement rate in psychotherapy is generally regarded as 50%, while 10% of clients deteriorate after therapy. This indicates a potential for improvement. Research shows that in therapies with the lack of progress, the clients rarely express dissatisfaction about progress to their therapists, and parallel, these therapists consider the therapies to proceed in the right direction. There is therefore a need for more knowledge about (a) how to obtain reliable information about the therapy progress and process monitored frequently during the course of therapy, and (b) that this information is fed back to the therapist and the client so that they (c) jointly can evaluate and adjust the aims and means for improving the therapy, something that may (d) enable them to test more appropriate approaches. This clinical practice should also enhance the client collaboration and empowerment in therapy, hopefully leading to higher recovery rate, shorter treatments, and reduced drop-out. To date, there is limited research on whether and how the use of feedback can contribute to improved outcomes. Such research is especially lacking in couple and family therapy. In a 3-year Norwegian pilot project at the Center for Family and relationships, Modum Bad, Department of Child and Adolescent Mental Health, Sørlandet Sykehus, and at Ålesund family counseling office, the online-based feedback system STIC (Systemic Therapy Inventory of Change) has been implemented and tested. The clinical experience is positive, and the system is considered suitable. This project has evolved parallel to a similar project at the Family Institute at Northwestern University, Evanston, Ill., supervised by the founder of the STIC system, professor William M. Pinsof. The project now enters a new phase by conducting a randomized, controlled trial (RCT) at three Norwegian couple- and family therapy sites in collaboration with five American psychotherapy sites to investigate whether the use of ongoing feedback is associated to more effective therapy compared with therapy without use of feedback.

ELIGIBILITY:
Inclusion Criteria:

* individuals,
* couples,
* families in Norwegian couple- and family therapy contexts

Exclusion Criteria:

* psychosis,
* current drug and alcohol abuse,
* violent and threatening behavior,
* not enable to understand Norwegian or English language.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KariAnne Vrabel, PhD, Study Director — Modum Bad Research Institute
Locations (3):
- Norway (3):
  - Drammen - Kongsberg family agency, Drammen, Buskerud
  - Center for family and relationship, Modum Bad, Vikersund, Buskerud
  - ABUP, Sørlandet sykehus, Kristiansand, Vest Agder

REFERENCES:
- [Background] Pinsof WM, Zinbarg RE, Lebow JL, Knobloch-Fedders LM, Durbin E, Chambers A, Latta T, Karam E, Goldsmith J, Friedman G. Laying the foundation for progress research in family, couple, and individual therapy: the development and psychometric features of the initial systemic therapy inventory of change. Psychother Res. 2009 Mar;19(2):143-56. doi: 10.1080/10503300802669973. PMID 19235092
- [Derived] Tilden T, Johnson SU, Hoffart A, Zahl-Olsen R, Wampold BE, Ulvenes P, Haland AT. Alliance predicting progress in couple therapy. Psychotherapy (Chic). 2021 Sep;58(3):391-400. doi: 10.1037/pst0000355. Epub 2021 Feb 4. PMID 33539145
- See also: Presentation of the Psychotherapy Change Project which is the overarching project for the STIC system. — http://www.family-institute.org/research/dan-j-epstein-family-foundation-center-for-psychotherapy-change

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected from 2013 to 2016 from three couple and family therapy sites in Norway.
Groups:
- The Use of STIC Feedback System: This condition included the use of the STIC feedback system. This implied that before every therapy session clients completed the STIC questionnaire that was processed into a report that was sent to the client's therapist. He or she used this report to prepare for the session, for instance investigating whether treatment progress and process developed satisfactory, and whether there was a need to address topics mentioned in the report. Sharing the results with the client enabled the client to interpret his or her own results and as such user involvement was strengthened.
- Treatment as Usual: This condition did not include the use of the STIC feedback system, in other words, treatment as usual (TAU).
Period: Overall Study
Arm/Group | The Use of STIC Feedback System | Treatment as Usual
Started | 165 | 163
Completed | 97 | 87
Not Completed | 68 | 76
Not completed — Lost to Follow-up | 68 | 76

BASELINE CHARACTERISTICS:
Groups:
- The Use of STIC Feedback System: This condition included the use of the STIC feedback system.
- Treatment as Usual: This condition did not include the use of the STIC feedback system.
- Total: Total of all reporting groups
Arm/Group | The Use of STIC Feedback System | Treatment as Usual | Total
Number analyzed (Participants) | 165 | 163 | 328
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.28 (9.73) | 39.47 (8.63) | 39.86 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 79 | 77 | 156
Beck Depression Inventory [Mean (Standard Deviation); unit: Unit on a scale] — The Beck Depression Inventory (BDI-II - Beck et al., 1995a) is a widely used 21-item self-report questionnaire assessing cognitive, affective, motivational, and physiological symptoms of depression and variation over time. Items are scored on a scale from 0 to 3 and the sum-score expressed the depth of the depression, graded from no clinical depression (0-9), through mild (10-19), moderate (20-29) and severe depression (30-63). Population: The reason why the row number differs from the overall number is that some participants were still in treatment and/or did not reply at the end of data collection. Those reported here have delivered complete sets of data.
  Unit on a scale
    number analyzed (Participants) | 92 | 84 | 176
    (all) | 15.10 (11.38) | 16.02 (11.56) | 15.36 (11.47)

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory II
Description: The Beck Depression Inventory (BDI-II - Beck et al., 1995a) is a widely used 21-item self-report questionnaire assessing cognitive, affective, motivational, and physiological symptoms of depression and variation over time. Items are scored on a scale from 0 to 3 and the sum-score expressed the depth of the depression, graded from no clinical depression (0-9), through mild (10-19), moderate (20-29) and severe depression (30-63). The BDI shows adequate psychometric properties (Beck et al., 1995b).
Time Frame: The BDI was completed at the start and end of treatment. In this study the treatment length varied from two to 22 sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Use of STIC Feedback System | Treatment as Usual
Number analyzed (Participants) | 92 | 84
score on a scale
  Start of treatment | 15.10 (11.38) | 16.02 (11.56)
  End of treatment | 10.78 (11.28) | 9.35 (10.58)
Statistical Analysis 1: Comparison: The Use of STIC Feedback System vs Treatment as Usual; Test type: Other — The BDI's Cronbach's alpha was .93 at start of therapy, and .95 at the end of therapy; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 1.01

ADVERSE EVENTS:
Time Frame: During treatment that varied from two to 22 sessions, with an average of four months.
Description: This was a non-invasive study where participants responded to standardized questionnaires. For this reason we hypothesize that there was no risk of mortality or serious adverse events caused by this study participation.
Arm/Group | The Use of STIC Feedback System | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/163
Other Adverse Events (participants affected / at risk) | 5/165 | 3/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Use of STIC Feedback System (N=165) | Treatment as Usual (N=163)
Stressor (Social circumstances) | 0 (0) | 0 (0) — Participating in the study could possibly increase the stress for the participants as completing questionniares added to their general life stress at the moment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | The Use of STIC Feedback System (N=165) | Treatment as Usual (N=163)
Clients felt that data collection was a burden (Investigations) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No